CLINICAL TRIAL: NCT00293098
Title: Compassionate Use of Deferiprone in Patients With Thalassemia and Iron-Induced Heart Disease
Brief Title: Compassionate Use of Deferiprone for Patients With Thalassemia and Iron-Induced Heart Disease
Status: Approved for marketing | Type: Expanded Access
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: ApoPharma (Industry)
Responsible Party: Principal Investigator, Alan Cohen, Chair, Department of Pediatrics, Children's Hospital of Philadelphia
Other Study IDs: 2006-2-4700
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Iron Overload
Keywords: Iron overload; Thalassemia; Iron induced heart disease; deferoxamine (Desferal); Deferiprone
MeSH Terms: conditions — Iron Overload; Thalassemia | interventions — Deferiprone

INTERVENTIONS:
Drug: deferiprone — oral administration of 75 mg/kg/day in three divided doses, usually in combination with deferoxamine therapy
  Other Names: Ferriprox

SUMMARY:
Patients who have iron overload due to chronic blood transfusions and have developed heart failure or who are at high risk of heart failure because of the high levels of iron in their hearts, will be treated with deferiprone, an investigational drug, in combination with deferoxamine (Desferal). Some studies suggest that deferiprone may be better than deferoxamine in removing iron from the heart and improving heart function, and that using both drugs together may remove more iron. Participants would make a clinic visit for lab studies each week, and would continue to take deferiprone for as long as their physician feels it is useful in their care.

DETAILED DESCRIPTION:
Repeated red cell transfusions lead to transfusional iron overload because the body lacks an efficient mechanism to excrete excess iron. Without treatment, iron accumulates in the liver, heart and endocrine glands. Cardiac complications including arrhythmias and congestive heart failure are the most common cause of death from transfusional iron overload. New magnetic resonance imaging (MRI) T2* techniques enable an estimation of cardiac iron loading, and allow patients at the highest risk of cardiac disease (those with T2* < 10 ms) to be identified. For over 30 years, deferoxamine has been the standard therapy. However, the mode of administration is cumbersome (subcutaneous or intravenous infusion over 8 to 12 hours daily), leading to poor compliance. Thus, cardiac disease and early mortality continue to be a significant problem in patients treated with chronic transfusions. Treatment of cardiac complications involves intensifying therapy with deferoxamine, including recommending intravenous administration over a period of 24 hours daily. Deferiprone is an oral chelating agent, not FDA approved for use in the United States. Recent studies indicate that deferiprone is superior to deferoxamine in removing cardiac iron and reducing iron-induced cardiotoxicity. The most serious side effect of deferiprone is agranulocytosis, and other side effects are gastrointestinal symptoms, reversible arthralgia, reddish discoloration of urine and rare cases of autoimmune disease. Patients on the study will be closely monitored for these toxicities. Patients who are currently regularly followed at The Children's Hospital of Philadelphia will be prescribed deferiprone at 75 mg/kg/day in three divided doses, taken orally, in combination with deferoxamine, at the patient's current dose. Labs will be drawn once per week to monitor neutrophil count, with additional labs every three months to monitor ferritin and ALT levels.

ELIGIBILITY:
Inclusion Criteria:

* Transfusional iron overload
* Overt cardiac failure or significant arrhythmia, OR high risk of developing cardiac failure as determined by T2* < 10 ms by magnetic resonance imaging (MRI)
* Signed consent form
* Patient regularly followed at The Children's Hospital of Philadelphia
* Unwillingness to participate in, or lack of suitability for, a clinical trial providing similar therapy

Exclusion Criteria:

* Previously treated with deferiprone and had severe adverse reactions necessitating discontinuation
* Receiving other investigational drugs
* Receiving other drugs known to cause neutropenia
* Unexplained occurrences of neutropenia in past two years
* Pregnant or breastfeeding; or want to become pregnant.
* Sexually active but unwilling to use reliable birth control
* Other conditions which, in the opinion of the investigator, would make patient unsuitable for enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Cohen, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States